CLINICAL TRIAL: NCT03593044
Title: Side Effects of Atropine (SEA) Study
Acronym: SEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeffrey J. Walline, OD PhD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey J. Walline, OD PhD, Associate Dean For Research, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0224
Record Dates: First submitted 2018-06-27; First posted 2018-07-19 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Myopia
Keywords: atropine; photophobia; pupil; reading speed; myopia; Surveys and Questionnaires
MeSH Terms: conditions — Myopia; Photophobia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Subjects will take drops for one week and measurements will be taken before and after treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- One Week Atropine (Experimental): 0.01% concentration atropine drops
  Interventions: Drug: 0.01% concentration atropine drops

INTERVENTIONS:
Drug: 0.01% concentration atropine drops — One drop of 0.01% concentration atropine in each eye at night for seven days.
  Other Names: Atropine Sulfate

SUMMARY:
This study will perform several objective and subjective measurements of the eye and vision before and after a week of using 0.01% concentration atropine drops. These measurements will help to obtain a comprehensive understanding of the side effects of this concentration of atropine and determine if the drops would be tolerated as a possible preventative treatment for nearsightedness.

DETAILED DESCRIPTION:
Atropine drops are commonly used to dilate the eye and prevent the ability to focus and also slow the progression of nearsightedness. Low concentration (0.01%) atropine slows the progression of myopia 60% to 83% while causing less side effects than high concentration (1.0%) atropine though still showing an effect on pupil size and pupil response.This study is a prospective cohort study in which several objective and subjective measurements will be taken before and after the use of 0.01% atropine for a week to determine the effect of this concentration on 1. vision at distance and near; 2. pupil size; 3. focusing ability, accuracy, and change; 4. symptoms, including subjective vision, headaches, light sensitivity, drop comfort; and 5. pressure in the eye. This will allow us to determine the effect these drops have on the eye and whether or not patients would be willing to use them as a possible preventative treatment for nearsightedness. The investigators expect to find that the drops will not affect vision, will increase pupil size, decrease focusing ability and accuracy (but not clinically meaningfully), cause some light sensitivity, and have no effect on eye pressure. The investigators expect that patients would be willing to use these drops to control nearsightedness even after experiencing the side effects.

ELIGIBILITY:
Inclusion Criteria:

-N/A

Exclusion Criteria:

* Outside of age range
* History of accommodative (focusing) issues or therapy

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Walline, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Clark TY, Clark RA. Atropine 0.01% Eyedrops Significantly Reduce the Progression of Childhood Myopia. J Ocul Pharmacol Ther. 2015 Nov;31(9):541-5. doi: 10.1089/jop.2015.0043. Epub 2015 Jul 28. PMID 26218150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects aged 22 to 26 years were enrolled in the study from July 2018 to January 2019.
Period: Overall Study
Arm/Group | One Week Atropine
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Spherical equivalent manifest refraction [Mean (Standard Deviation); unit: diopters] — The spherical equivalent manifest refraction equals the spherical component of the manifest refraction plus one-half of the cylinder component (astigmatism) of the manifest refraction. This is a measure of the refractive error (near-sightedness or far-sightedness) of the subject's eye and is performed using an instrument called a phoropter with multiple lenses of differing powers to investigate which lens makes the patient's vision look the clearest.
  diopters | -3.12 (2.87)
Eye color [Count of Participants; unit: Participants]
  Brown | 12
  Blue | 11
  Green | 7
  Hazel | 1

OUTCOME MEASURES:

1. Primary Outcome: Diameter of the Pupil Measured With a Neuroptix Pupillometer
Description: Change in pupil size between baseline visit and follow up visit (after one week on treatment) in millimeters to the nearest tenth of a millimeter
Time Frame: Baseline (before) and one week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
millimeters
  Photopic pupil size before administration of drops | 4.9 (0.8)
  Photopic pupil size after administration of drops for one week | 5.1 (0.6)
  Mesopic pupil size before administration of drops | 5.9 (0.66)
  Mesopic pupil size after administration of drops for one week | 5.9 (0.7)
Statistical Analysis 1: Comparison: One Week Atropine; Photopic pupil size; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: One Week Atropine; Mesopic pupil size; Test type: Other; p = 0.66, t-test, 2 sided

2. Primary Outcome: Visual Acuity With Bailey-Lovie logMAR Visual Acuity Charts
Description: Investigators will measure the change in high contrast distance and near logMAR visual acuity and low contrast distance logMAR visual acuity between baseline visit and follow up visit (after one week on treatment).
Time Frame: Baseline (before) and one week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
logMAR
  High contrast distance visual acuity before drops | -0.1 (0.1)
  High contrast distance visual acuity after administration of drops for one week | -0.1 (0.1)
  High contrast near visual acuity before drops | -0.2 (0.1)
  High contrast near visual acuity adter administration of drops for one week | -0.2 (0.1)
  Low contrast visual acuity before drops | 0.0 (0.1)
  Low contrast visual acuity after administration of drops for one week | 0.0 (0.1)
Statistical Analysis 1: Comparison: One Week Atropine; High contrast distance visual acuity; Test type: Other; p = 0.96, t-test, 2 sided
Statistical Analysis 2: Comparison: One Week Atropine; High contrast near visual acuity; Test type: Other; p = 0.77, t-test, 2 sided
Statistical Analysis 3: Comparison: One Week Atropine; Low contrast distance visual acuity; Test type: Other; p = 0.82, t-test, 2 sided

3. Secondary Outcome: Eye Focusing Measured by the Closest One Can Read a Letter and Focusing Accuracy Measured by an Autorefractor
Description: Investigators will measure the change in near point of accommodation (how close an object can be seen clearly) in centimeters and accommodative lag (error of focusing on near objects) in diopters.
Time Frame: One week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
diopters
  Accommodative amplitude before drops | 8.1 (1.2)
  Accommodative amplitude after administration of drops for one week | 8.5 (1.3)
  Accommodative lag before drops | -0.8 (1.7)
  Accommodative lag after administration of drops for one week | -0.9 (0.8)
  Accommodative facility before drops | 13.6 (4)
  Accommodative facility after administration of drops for one week | 14.0 (3.8)
Statistical Analysis 1: Comparison: One Week Atropine; Accommodative amplitude; Test type: Other; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: One Week Atropine; Accommodative lag; Test type: Other; p = 0.66, t-test, 2 sided
Statistical Analysis 3: Comparison: One Week Atropine; Accommodative facility; Test type: Other; p = 0.24, t-test, 2 sided

4. Secondary Outcome: Change in Subjective Assessment of Potential Side Effects by Asking the Same Questions Before and After Administration of Eye Drops.
Description: Each of the below scores are from an individual question that was answered before taking atropine drops and after taking atropine drops nightly for one week.
  Glare: 1 (good) to 10 (perfect); 10 is best Ghost images: 1 (good) to 10 (perfect); 10 is best Straing/tiredness: 1 (good) to 10 (perfect); 10 is best Changing vision: 1 (good) to 10 (perfect); 10 is best Headache frequency: 1 (very infrequent) to 10 (very frequent); 1 is best Distance clarity: 1 (good) to 10 (perfect): 10 is best Computer clarity: 1 (good) to 10 (perfect); 10 is best Small print clarity: 1 (good) to 10 (perfect); 10 is best Sports/hobbies vision: 1 (good) to 10 (perfect); 10 is best Overall vision: 1 (good) to 10 (perfect); 10 is best Light sensitivity: 1 (not sensitive at all) to 10 (very sensitive); 10 is best Discomfort during bright light: 1 (no discomfort) to 10 (extreme discomfort); 1 is best
Time Frame: Baseline (before) and one week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: score on a question from 1 to 10
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
score on a question from 1 to 10
  Glare before drops | 8.7 (1.9)
  Glare after drops | 9.0 (1.3)
  Ghost images before drops | 9.8 (0.9)
  Ghost images after drops | 9.7 (0.7)
  Strain/tiredness before drops | 8.3 (1.5)
  strain/tiredness after drops | 8.7 (1.6)
  Changing vision before drops | 9.4 (1.2)
  Changing vision after drops | 9.4 (0.9)
  Headache frequency before drops | 1.6 (0.5)
  Headache frequency after drops | 1.7 (0.5)
  Distance clarity before drops | 8.8 (1.5)
  Distance clarity after drops | 8.7 (1.2)
  Computer clarity before drops | 9.5 (0.8)
  Computer clarity after drops | 9.3 (1.0)
  Small print clarity before drops | 9.5 (1.1)
  Small print clarity after drops | 9.1 (1.0)
  Vision during sports/hobbies before drops | 9.6 (0.6)
  Vision during sports/hobbies after drops | 9.6 (0.6)
  Overall vision before drops | 9.4 (1.0)
  Overall vision after drops | 9.1 (0.9)
  Light sensitivity before drops | 2.8 (2.5)
  Light sensitivity after drops | 3.1 (2.5)
  Discomfort during bright light before drops | 2.7 (1.9)
  Discomfort during bright light after drops | 2.0 (1.7)
Statistical Analysis 1: Comparison: One Week Atropine; Glare; Test type: Other; p = 0.3, t-test, 2 sided
Statistical Analysis 2: Comparison: One Week Atropine; Ghost images; Test type: Other; p = 0.5, t-test, 2 sided
Statistical Analysis 3: Comparison: One Week Atropine; Strain/tiredness; Test type: Other; p = 0.9, t-test, 2 sided
Statistical Analysis 4: Comparison: One Week Atropine; Changing vision; Test type: Other; p = 0.9, t-test, 2 sided
Statistical Analysis 5: Comparison: One Week Atropine; Headache frequency; Test type: Other; p = 0.3, t-test, 2 sided
Statistical Analysis 6: Comparison: One Week Atropine; Distance clarity; Test type: Other; p = 0.7, t-test, 2 sided
Statistical Analysis 7: Comparison: One Week Atropine; Computer clarity; Test type: Other; p = 0.3, t-test, 2 sided
Statistical Analysis 8: Comparison: One Week Atropine; Small print clarity; Test type: Other; p = 0.1, t-test, 2 sided
Statistical Analysis 9: Comparison: One Week Atropine; Vision during sports/hobbies; Test type: Other; p = 1.0, t-test, 2 sided
Statistical Analysis 10: Comparison: One Week Atropine; Overall vision; Test type: Other; p = 0.2, t-test, 2 sided
Statistical Analysis 11: Comparison: One Week Atropine; Light sensitivity; Test type: Other; p = 0.7, t-test, 2 sided
Statistical Analysis 12: Comparison: One Week Atropine; Discomfort during bright light; Test type: Other; p = 0.002, t-test, 2 sided

5. Secondary Outcome: Change in Intraocular Pressure Using a Tonopen
Description: We will measure the change in eye pressure between baseline visit and follow up visit (after one week on treatment) measured with Tonopen and recorded in mmHg.
Time Frame: Baseline (before) and one week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: millimeters Mercury
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
millimeters Mercury
  Intraocular pressure of right eyes before drops | 15.5 (2.9)
  Intraocular pressure of right eyes after administration of drops for one week | 17.0 (2.8)
  Intraocular pressure of left eyes before drops | 15.7 (2.8)
  Intraocular pressure of left eyes after administration of drops for one week | 16.4 (3.1)
Statistical Analysis 1: Comparison: One Week Atropine; Right eye intraocular pressure; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: One Week Atropine; Left eye intraocular pressure; Test type: Other; p = 0.05, t-test, 2 sided

6. Secondary Outcome: Ability to Change Focus From Far to Near Measured by Stimulating and Relaxing Focus of the Eyes as Many Times as Possible in One Minute.
Description: Investigators will measure accommodative facility (ability to change focus from far to near) in number of cycles between baseline visit and follow up visit (after one week on treatment).
Time Frame: Baseline (before) and one week after beginning treatment with drops
Measure: Mean (Standard Deviation); unit: cycles per minute
Arm/Group | One Week Atropine
Number analyzed (Participants) | 31
cycles per minute
  Accommodative facility before drops | 13.6 (4)
  Accommodative facility after administering drops for one week | 14.0 (3.8)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | One Week Atropine
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03593044/Prot_SAP_002.pdf
  • Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03593044/ICF_004.pdf